CLINICAL TRIAL: NCT01262222
Title: Endothelial Dysfunction in Patients Undergoing Major Cancer Surgery: Incidence and Predictive Value for Postoperative Cardiac Events
Brief Title: Patients Undergoing Major Cancer Surgery: Incidence and Predictive Value for Postoperative Cardiac Events
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-206
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: High Risk for Postoperative Cardiovascular Events
Keywords: Predictive Value For Postoperative Cardiac Events; Endothelial Dysfunction; 10-206

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood draw

GROUPS / COHORTS (1):
- pts undergoing major surg procedure referred to cardiology: Patients deemed to be at intermediate to high risk for postoperative cardiovascular events by clinical criteria will be the subject of this study. Cardiac risk will be determined according to the Revised Cardiac Risk Index (RCRI). RH-PAT testing and BNP evaluation will take place within 30 days before surgery and may occur on separate days. The blood may be drawn on the day of the RH-PAT testing or at a time of routine blood drawing within the 30 day period. After surgery the patient will be monitored and examined in the PACU for evidence of cardiac events.
  Interventions: Other: endothelial function testing

INTERVENTIONS:
Other: endothelial function testing — After obtaining informed consent, eligible patients will undergo endothelial function testing using the Endo-PAT 2000 (Itamar Medical) device. This PAT device applied to the finger tip will be used to measure change in blood flow in one arm at rest and after a 5 minute occlusion of the brachial artery with a blood pressure cuff. The other arm will serve as the patient's own control. After the cuff is deflated, blood flow normally increases in the arm for a period of time (flow mediated dilatation). In patients with abnormal endothelial function, this increase in blood flow is damped. The ratio of flow in the ischemic finger to the nonischemic finger (RH-PAT) will then be correlated with postoperative cardiac events.

SUMMARY:
The purpose of this study is to look at a new method for finding out if patients have a risk of heart complications from surgery. At the present, to find out if patients have a risk of heart complications from surgery, look at whether the patient has heart disease, diabetes, kidney problems, and stroke. The investigators hope that this study will confirm a new, safe test to help us predict the risk of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Undergoing High Risk Cancer Surgery (Patient must be undergoing one of the following procedures NOTE: All open or robotic forms of the following procedures meet the eligibility criteria. GMT/ Hepatobiliary
* Pancreatic Resection
* Retroperitoneal Sarcomas
* Shoulder (Forequarter) Amputation
* Esophagectomy, Esophagogastrectomy
* Pheochromocytoma
* Liver Resection (with or without Bile Duct Resection) Orthopedics
* Spine Resections (with or without Spinal Fusion)
* Metastatic Disease Requiring Total Hip Replacement
* Total Shoulder Replacement / Forequarter Amputation
* Hemipelvectomy
* Sacrectomy Thoracic
* Extrapleural Pneumonectomy
* Pleurectomy and Decortication
* Pneumonectomy
* Esophagogastrectomy
* Mediastinal Tumor Resection
* Pancoast Tumor
* Completion Pneumonectomy
* Lobectomy (post-induction chemotherapy; or severe COPD)
* Segmentectomy Colorectal/ GYN
* Colon Resection with possible Sacrectomy
* Pelvic Exenteration
* Advanced ovarian cancer resection with or without liver resection Urology
* Radical Cystectomy
* Open Radical Prostatectomy
* Nephrectomy with Vena Caval Resection Head & Neck
* Thyroid Resection with Mediastinal involvement
* Major head and neck cancer resection with Free Flap reconstruction Other
* Unclassified Major Surgery at the Discretion of the PI
* Postoperative stay likely to be 2 or more days
* Patients willing to tolerate inflation of a blood pressure cuff for 5 minutes
* Patients willing to cut long nails in order to wear finger probe.
* Patients with one or more of the following RCRI risk factors:
* History of ischemic heart disease (any)
* History of myocardial infarction
* History of positive exercise test
* Current complaint of chest pain considered secondary to myocardial ischemia
* Use of nitrate therapy
* ECG with pathological Q waves
* History of congestive heart failure (any)
* History of congestive heart failure
* Pulmonary edema
* Paroxysmal nocturnal dyspnea
* Bilateral rales or S3 gallop
* Chest radiograph showing pulmonary vascular redistribution
* History of cerebrovascular disease (any)
* History of transient ischemic attack (TIA) or stroke
* Preoperative treatment with insulin
* Preoperative serum creatinine > 2.0 mg/dL
* Evidence of peripheral vascular disease other than cerebral vascular disease (Although peripheral vascular disease is not strictly a RCRI risk factor, Fleisher indicates: "It would not be inappropriate to assume that any atherosclerotic class of disease is equivalent to ischemic heart disease for risk purposes."

Exclusion Criteria:

* Medical conditions precluding use of arm blood pressure measurements such as prior lymphadenectomy, vascular shunts for dialysis or upper extremity occlusive vascular disease
* Patients undergoing emergency surgery
* Any of the following active conditions
* Unstable coronary syndromes
* Uncompensated heart failure; worsening or new onset CHF
* Significant arrhythmias
* Atrial fibrillation, presently
* High grade AV block
* Symptomatic ventricular arrhythmias or new ventricular arrhythmias
* Supraventricular arrhythmias with poor rate control
* Symptomatic bradycardia
* Severe valvular disease
* Severe aortic stenosis (mean transvalvular gradient >40mmHg)
* Symptomatic mitral stenosis
* Any other condition that at the judgment of the investigator might require additional evaluation and treatment before surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for major intrathoracic or intraabdominal surgery who meet inclusion criteria and are seen either in preoperative cardiology consultation or by another pre-surgical service such as general medicine will be eligible for screening.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2010-12; Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
To determine whether endothelial dysfunction as measured by abnormal flow mediated dilation (FMD). | 1 year
  Identifies patients at high risk of cardiovascular complications after major thoracic or abdominal cancer surgery.

SECONDARY OUTCOMES:
To obtain preliminary information on whether abnormal FMD adds predictive information beyond risk algorithms | 1 year
  proposed by the American Heart Association/American College of Cardiology.
To determine whether abnormal flow mediated dilation (FMD) correlates to abnormal brain natriuretic enzyme BNP levels prior to surgery. | 1 year
To survey whether FMD prior to surgery is affected by treatment with chemotherapy and/or radiation prior to major cancer surgery | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm